CLINICAL TRIAL: NCT00771030
Title: A Randomized, Double-blind, Placebo-controlled, Ascending Multiple-dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Efficacy of AMG 827 in Subjects With Rheumatoid Arthritis
Brief Title: Study to Evaluate the Safety, PK, PD and Efficacy of AMG 827 in Adults With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20070264
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Results first posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — brodalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (7):
- Placebo SC (Cohorts 1-3) (Placebo Comparator): Participants received placebo to brodalumab by subcutaneous (SC) injection once every 2 weeks for a total of six doses.
  Interventions: Other: Placebo
- Placebo IV (Cohorts 5-6) (Placebo Comparator): Participants received placebo to brodalumab by intravenous (IV) infusion every 4 weeks for a total of two doses.
  Interventions: Other: Placebo
- Brodalumab 50 mg SC (Cohort 1) (Experimental): Participants received 50 mg brodalumab by subcutaneous injection once every 2 weeks for a total of six doses.
  Interventions: Biological: Brodalumab
- Brodalumab 140 mg SC (Cohort 2) (Experimental): Participants received 140 mg brodalumab by subcutaneous injection once every 2 weeks for a total of six doses.
  Interventions: Biological: Brodalumab
- Brodalumab 210 mg SC (Cohort 3) (Experimental): Participants received 210 mg brodalumab by subcutaneous injection once every 2 weeks for a total of six doses.
  Interventions: Biological: Brodalumab
- Brodalumab 420 mg IV (Cohort 5) (Experimental): Participants received 420 mg brodalumab by IV infusion once every 4 weeks for a total of two doses.
  Interventions: Biological: Brodalumab
- Brodalumab 700 mg IV (Cohort 6) (Experimental): Participants received 700 mg brodalumab by IV infusion once every 4 weeks for a total of two doses.
  Interventions: Biological: Brodalumab

INTERVENTIONS:
Biological: Brodalumab — Solution for subcutaneous or intravenous administration
  Other Names: AMG 827
  Arms: Brodalumab 140 mg SC (Cohort 2); Brodalumab 210 mg SC (Cohort 3); Brodalumab 420 mg IV (Cohort 5); Brodalumab 50 mg SC (Cohort 1); Brodalumab 700 mg IV (Cohort 6)
Other: Placebo — Solution for subcutaneous or intravenous administration
  Arms: Placebo IV (Cohorts 5-6); Placebo SC (Cohorts 1-3)

SUMMARY:
This Phase 1b/2a study will evaluate safety, tolerability pharmacokinetics (PK) and pharmacodynamics (PD) of brodalumab when administered in multiple subcutaneous (SC) and intravenous (IV) doses in patients with active rheumatoid arthritis (RA) in combination with a stable dose of disease modulating anti-rheumatic drugs (DMARDs). Part A is dose escalation (to assess safety & tolerability), and Part B is dose expansion (to assess clinical efficacy) at the highest tolerated dose level of brodalumab from Part A.

DETAILED DESCRIPTION:
The dose-escalation phase consisted of 5 sequentially enrolled dose cohorts. Within each cohort participants were randomly assigned in a 3:1 ratio to receive brodalumab or placebo subcutaneously (cohorts 1 to 3) or intravenously (cohorts 5 and 6).

Dose escalations required acceptable safety data based on blinded review following completion of the day 15/week 3 visit by the final participant in each cohort and when six or more participants in a cohort had been administered at least three doses of brodalumab (cohorts 1, 2, 3 and 5). In cohort 6, dose escalation followed completion of the day 15/week 3 visit by the final patient in cohort 5 and six or more participants in cohort 5 had been administered two or more IV infusions of brodalumab.

Cohort 4 was designed to be used in the dose expansion phase to provide evidence of biological impact in 70 patients with RA receiving brodalumab at the dose determined during the dose escalation phase of the study. This cohort was not enrolled because a decision was made not to conduct Part B of the study; instead a separate phase 2 multiple-dose study was conducted to evaluate efficacy of brodalumab in patients with RA (Study 20090061; NCT00950989).

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 to 70 years of age, inclusive at the time of screening
* Diagnosed with RA as determined by meeting 1987 American College of Rheumatology (ACR) classification criteria
* Active RA defined as ≥ 6 swollen joints (out of 66 joints examined) and ≥ 8 tender/painful joints (out of 68 joints examined) and at least 1 of the following:
* Erythrocyte sedimentation rate (ESR) ≥ 28 mm, or
* C-reactive protein (CRP) > 15 mg/L, or
* Morning stiffness > 45 minutes (applicable to subjects in Part A ONLY)
* Duration of RA for at least 6 months
* Currently taking methotrexate (MTX) consecutively for ≥ 12 weeks and on a stable dose of oral or SC MTX at 15-25 mg weekly for ≥ 4 weeks at day -1. A lower MTX dose is acceptable if it is the highest tolerated dose, however, toxicity documentation by the Investigator is required. All subjects will take folic acid to minimize toxicity, according to local guidelines.
* Additional Inclusion Criteria Apply

Exclusion Criteria:

* History or evidence of a clinically significant disorder other than RA (including but not limited to cardiopulmonary, oncologic, renal, metabolic, hematologic or psychiatric), condition or disease that, in the opinion of the Investigator and Amgen physician would pose a risk to subject safety or interfere with the study evaluation, procedures or completion
* Uncontrolled, clinically significant systemic disease other than RA such as diabetes mellitus, liver disease, asthma, cardiovascular disease or hypertension
* Malignancy within 5 years (except successfully treated in situ cervical cancer or squamous or basal cell carcinoma of the skin)
* Presence of a serious or chronic infections
* Subject (male or female) is not willing to use highly effective contraception, defined as a double barrier method (ie, spermicidal jelly and condom, or condom and diaphragm) during treatment and up to end of study
* Additional Exclusion Criteria Apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-10-27 (Actual); Primary Completion 2010-05-25 (Actual); Study Completion 2010-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Martin DA, Churchill M, Flores-Suarez L, Cardiel MH, Wallace D, Martin R, Phillips K, Kaine JL, Dong H, Salinger D, Stevens E, Russell CB, Chung JB. A phase Ib multiple ascending dose study evaluating safety, pharmacokinetics, and early clinical response of brodalumab, a human anti-IL-17R antibody, in methotrexate-resistant rheumatoid arthritis. Arthritis Res Ther. 2013 Oct 25;15(5):R164. doi: 10.1186/ar4347. PMID 24286136
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 11 sites: 7 in the United States, 2 in Canada and 2 in Mexico.
Pre-assignment Details: Within each cohort participants were randomized 3:1 to receive ascending doses of brodalumab or placebo subcutaneously (cohorts 1 to 3) or intravenously (cohorts 5 and 6).
  Cohort 4 was designed to be used in the dose expansion part of the study, however, this cohort was not enrolled because experimental endpoints would be achieved during a separate phase II study.
Period: Overall Study
Arm/Group | Placebo SC (Cohorts 1-3) | Placebo IV (Cohorts 5-6) | Brodalumab 50 mg SC (Cohort 1) | Brodalumab 140 mg SC (Cohort 2) | Brodalumab 210 mg SC (Cohort 3) | Brodalumab 420 mg IV (Cohort 5) | Brodalumab 700 mg IV (Cohort 6)
Started | 6 | 4 | 6 | 6 | 6 | 6 | 6
Received Study Drug (Study drug refers to placebo or brodalumab) | 6 | 4 | 6 | 6 | 6 | 6 | 6
Completed | 6 | 3 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo SC (Cohorts 1-3) | Placebo IV (Cohorts 5-6) | Brodalumab 50 mg SC (Cohort 1) | Brodalumab 140 mg SC (Cohort 2) | Brodalumab 210 mg SC (Cohort 3) | Brodalumab 420 mg IV (Cohort 5) | Brodalumab 700 mg IV (Cohort 6) | Total
Number analyzed (Participants) | 6 | 4 | 6 | 6 | 6 | 6 | 6 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (10.3) | 55.5 (11.7) | 46.2 (11.7) | 56.8 (8.7) | 45.7 (10.1) | 55.5 (7.3) | 50.0 (5.9) | 51.4 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 6 | 6 | 5 | 5 | 3 | 34
  Male | 1 | 0 | 0 | 0 | 1 | 1 | 3 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 2 | 3 | 2 | 1 | 5 | 1 | 18
  Black or African American | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Hispanic or Latino | 1 | 1 | 3 | 4 | 4 | 1 | 5 | 19
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment, including any such occurrence (eg, sign, symptom, or diagnosis) or worsening of a pre-existing medical condition.
  A serious adverse event was defined as an adverse event that was fatal; was life threatening; required in-patient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect; or other significant medical hazard.
Time Frame: From first dose of study drug up to end of study (week 19).
Population: All randomized participants who received at least 1 dose of study drug (placebo or brodalumab).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo SC (Cohorts 1-3) | Placebo IV (Cohorts 5-6) | Brodalumab 50 mg SC (Cohort 1) | Brodalumab 140 mg SC (Cohort 2) | Brodalumab 210 mg SC (Cohort 3) | Brodalumab 420 mg IV (Cohort 5) | Brodalumab 700 mg IV (Cohort 6)
Number analyzed (Participants) | 6 | 4 | 6 | 6 | 6 | 6 | 6
Participants
  Any treatment-emergent adverse event (TEAE) | 3 | 4 | 5 | 5 | 4 | 5 | 4
  Serious TEAEs | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Treatment-related TEAEs | 1 | 2 | 0 | 3 | 2 | 2 | 0
  Treatment-related serious TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Discontinuation of study drug due to TEAE | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Deaths on study | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Clinically Significant Changes in Safety Laboratory Tests
Description: The investigator reviewed laboratory test results and determined whether an abnormal value in an individual study participant represented a change from prestudy values and determined if changes were clinically significant. The number of participants with clinically significant changes in lab values at any time during the study is reported.
Time Frame: Blood samples were taken on days 2, 8, 15, 29, 43, 57, 71, 85, 106, and 127.
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo SC (Cohorts 1-3) | Placebo IV (Cohorts 5-6) | Brodalumab 50 mg SC (Cohort 1) | Brodalumab 140 mg SC (Cohort 2) | Brodalumab 210 mg SC (Cohort 3) | Brodalumab 420 mg IV (Cohort 5) | Brodalumab 700 mg IV (Cohort 6)
Number analyzed (Participants) | 6 | 4 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Changes in Physical Examination Findings, Vital Signs, or Electrocardiogram Findings
Time Frame: From first dose of study drug up to 4 weeks after last dose; 14 weeks for Cohorts 1, 2, and 3 and 8 weeks for Cohorts 5 and 6.
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo SC (Cohorts 1-3) | Placebo IV (Cohorts 5-6) | Brodalumab 50 mg SC (Cohort 1) | Brodalumab 140 mg SC (Cohort 2) | Brodalumab 210 mg SC (Cohort 3) | Brodalumab 420 mg IV (Cohort 5) | Brodalumab 700 mg IV (Cohort 6)
Number analyzed (Participants) | 6 | 4 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Anti-brodalumab Antibodies
Description: Samples were tested in a validated immunoassay for the presence of anti-brodalumab binding antibodies. Samples found to be positive for binding antibodies were further tested using a validated cell-based bioassay to determine if the antibodies were able to neutralize the activity of brodalumab.
Time Frame: Days 1 (pre-dose), 29 (pre-dose), 85, and 127
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo SC (Cohorts 1-3) | Placebo IV (Cohorts 5-6) | Brodalumab 50 mg SC (Cohort 1) | Brodalumab 140 mg SC (Cohort 2) | Brodalumab 210 mg SC (Cohort 3) | Brodalumab 420 mg IV (Cohort 5) | Brodalumab 700 mg IV (Cohort 6)
Number analyzed (Participants) | 6 | 4 | 6 | 6 | 6 | 6 | 6
Participants
  Binding antibodies | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Neutralizing antibodies | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Time to Maximum Concentration of Brodalumab After Single and Multiple Subcutaneous Doses
Time Frame: After first dose on days 1 (pre-dose and 4 hours post-dose), 2, 3, 5, 8, 11, and 15 (pre-dose), and after last dose on days 71 (pre-dose and 4 hours post-dose), 72, 73, 75, 78, 81, 85, 106 and 127.
Population: Participants who received subcutaneously administered brodalumab with available data
Measure: Median (Full Range); unit: days
Arm/Group | Brodalumab 50 mg SC (Cohort 1) | Brodalumab 140 mg SC (Cohort 2) | Brodalumab 210 mg SC (Cohort 3)
Number analyzed (Participants) | 6 | 6 | 6
days
  Day 1 (first dose) | 1.46 [0.18 to 2.00] | 3.96 [2.00 to 4.00] | 2.99 [0.97 to 4.00]
  Day 71 (last dose) | 2.00 [1.13 to 2.09] | 3.95 [1.93 to 4.07] | 4.00 [1.02 to 4.02]

6. Secondary Outcome: Maximum Concentration of Brodalumab After Single and Multiple Subcutaneous Doses
Time Frame: as for outcome 5
Population: Participants who received subcutaneously administered brodalumab with available data
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Brodalumab 50 mg SC (Cohort 1) | Brodalumab 140 mg SC (Cohort 2) | Brodalumab 210 mg SC (Cohort 3)
Number analyzed (Participants) | 6 | 6 | 6
μg/mL
  Day 1 (first dose) | 0.742 (0.522) | 5.67 (2.98) | 16.6 (8.97)
  Day 71 (last dose) | 1.35 (1.07) | 5.93 (5.15) | 18.4 (7.21)

7. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to the Time of the Final Quantifiable Sample (AUC0-t) for Brodalumab After Single and Multiple Subcutaneous Doses
Time Frame: as for outcome 5
Population: Participants who received subcutaneously administered brodalumab with available data
Measure: Mean (Standard Deviation); unit: days*μg/mL
Arm/Group | Brodalumab 50 mg SC (Cohort 1) | Brodalumab 140 mg SC (Cohort 2) | Brodalumab 210 mg SC (Cohort 3)
Number analyzed (Participants) | 6 | 6 | 6
days*μg/mL
  Day 1 (first dose) | 1.77 (1.61) | 37.6 (27.8) | 142 (67.3)
  Day 71 (last dose) | 4.13 (3.20) | 50.8 (51.5) | 191 (82.7)

8. Secondary Outcome: Accumulation Ratio for Brodalumab After Subcutaneous Dosing
Description: Accumulation was measured by AUC0-t, last dose / AUC0-t, first dose).
Time Frame: as for outcome 5
Population: Participants who received subcutaneously administered brodalumab with available data
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Brodalumab 50 mg SC (Cohort 1) | Brodalumab 140 mg SC (Cohort 2) | Brodalumab 210 mg SC (Cohort 3)
Number analyzed (Participants) | 6 | 6 | 6
ratio | 24.4 (51.4) | 1.3 (0.8) | 1.5 (0.6)

9. Secondary Outcome: Time to Maximum Concentration of Brodalumab After Single and Multiple Intravenous Doses
Time Frame: After first dose on days 1 (pre-dose and 0.5 and 4 hours post-dose), 2, 3, 5, 8, 11, and 15, and after last dose on days 29 (pre-dose and 0.5 and 4 hours post-dose), 30, 31, 33, 36, 39, 43, 57, 85, 106 and 127.
Population: Participants who received brodalumab by intravenous infusion with available data
Measure: Median (Full Range); unit: hours
Arm/Group | Brodalumab 420 mg IV (Cohort 5) | Brodalumab 700 mg IV (Cohort 6)
Number analyzed (Participants) | 6 | 6
hours
  Day 1 (first dose) | 4.07 [3.40 to 22.27] | 0.92 [0.82 to 1.53]
  Day 29 (last dose): number analyzed (Participants) | 6 | 5
  Day 29 (last dose) | 0.98 [0.77 to 4.02] | 0.83 [0.57 to 4.55]

10. Secondary Outcome: Maximum Concentration of Brodalumab After Single and Multiple Intravenous Doses
Time Frame: as for outcome 9
Population: Participants who received brodalumab by intravenous infusion with available data
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Brodalumab 420 mg IV (Cohort 5) | Brodalumab 700 mg IV (Cohort 6)
Number analyzed (Participants) | 6 | 6
μg/mL
  Day 1 (first dose) | 111 (19.2) | 240 (44.8)
  Day 29 (last dose): number analyzed (Participants) | 6 | 5
  Day 29 (last dose) | 127 (12.1) | 655 (949)

11. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to the Time of the Final Quantifiable Sample (AUC0-t) for Brodalumab After Single and Multiple Intravenous Doses
Time Frame: as for outcome 9
Population: Participants who received brodalumab by intravenous infusion with available data
Measure: Mean (Standard Deviation); unit: days*μg/mL
Arm/Group | Brodalumab 420 mg IV (Cohort 5) | Brodalumab 700 mg IV (Cohort 6)
Number analyzed (Participants) | 6 | 6
days*μg/mL
  Day 1 (first dose) | 831 (197) | 1840 (602)
  Day 29 (last dose): number analyzed (Participants) | 6 | 5
  Day 29 (last dose) | 951 (307) | 2230 (998)

12. Secondary Outcome: Accumulation Ratio for Brodalumab After Intravenous Dosing
Description: Accumulation was measured by AUC0-t, last dose / AUC0-t, first dose).
Time Frame: as for outcome 9
Population: Participants who received brodalumab by intravenous infusion with available data
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Brodalumab 420 mg IV (Cohort 5) | Brodalumab 700 mg IV (Cohort 6)
Number analyzed (Participants) | 6 | 5
ratio | 1.1 (0.2) | 1.2 (0.1)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to end of study (week 19).
Arm/Group | Placebo SC (Cohorts 1-3) | Placebo IV (Cohorts 5-6) | Brodalumab 50 mg SC (Cohort 1) | Brodalumab 140 mg SC (Cohort 2) | Brodalumab 210 mg SC (Cohort 3) | Brodalumab 420 mg IV (Cohort 5) | Brodalumab 700 mg IV (Cohort 6)
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/4 | 0/6 | 0/6 | 0/6 | 1/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/6 | 4/4 | 5/6 | 5/6 | 4/6 | 5/6 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo SC (Cohorts 1-3) (N=6) | Placebo IV (Cohorts 5-6) (N=4) | Brodalumab 50 mg SC (Cohort 1) (N=6) | Brodalumab 140 mg SC (Cohort 2) (N=6) | Brodalumab 210 mg SC (Cohort 3) (N=6) | Brodalumab 420 mg IV (Cohort 5) (N=6) | Brodalumab 700 mg IV (Cohort 6) (N=6)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Complicated migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo SC (Cohorts 1-3) (N=6) | Placebo IV (Cohorts 5-6) (N=4) | Brodalumab 50 mg SC (Cohort 1) (N=6) | Brodalumab 140 mg SC (Cohort 2) (N=6) | Brodalumab 210 mg SC (Cohort 3) (N=6) | Brodalumab 420 mg IV (Cohort 5) (N=6) | Brodalumab 700 mg IV (Cohort 6) (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Administration site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Injection site erythema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site haematoma (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Amoebiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eschar (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 1 | 1 | 2 | 2 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Affect lability (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breast cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Menstrual disorder (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.